CLINICAL TRIAL: NCT05503758
Title: Quantification of Different Lumbar Paravertebral Muscles Properties in Women Who Experienced Cesarean Delivery Under Different Types of Anaesthesia
Brief Title: Biomechanical Properties of the Lumbar Paravertebral Muscles
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Assistant Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Lumbar Paravertebral muscles
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-04

CONDITIONS: Lumbar Paravertebral Muscles

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: 9 participants have exposed to midline epidural anaesthesia for cesarean delivery.
  Interventions: Device: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)
- Group B: 22 participants have exposed to midline spinal anaesthesia for cesarean delivery.
  Interventions: Device: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)
- Group C: 10 participants underwent general anesthesia for cesarean delivery.
  Interventions: Device: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)
- Group D: 22 participants were in the control group (no previous pregnancy or anaesthesia).
  Interventions: Device: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia)

INTERVENTIONS:
Device: Myoton PRO device (MyotonPRO; Myoton AS, Tallinn, Estonia) — The MyotoPRO device is a portable objective device for measuring the contractile (tone), and biomechanical (stiffness) properties of lumbar paravertebral muscles (LPVMs).
  Other Names: Myotonometry

SUMMARY:
Cesarean delivery (CD) is an obstetric surgery for fetal delivery that involves both an abdominal incision (laparotomy) and a uterine incision (hysterotomy). It is presently the most prevalent surgery in the United States, with over 1 million women giving birth by cesarean section each year.

DETAILED DESCRIPTION:
The anaesthetic types of choice for cesarean delivery are neuraxial and general anaesthesia.

Neuraxial anesthesia is the gold standard anaesthesia for CD; it includes spinal and epidural anaesthesia. For spinal anaesthesia, local anesthetics are injected into the spinal canal, while for epidural anaesthesia, they are injected into the epidural space.

Despite the superiority of neuraxial anaesthesia for cesarean delivery, general anesthesia is still performed to some extent especially when neuraxial anaesthesia is failed or inconsistent.

General anesthesia involves a transient state of unconsciousness through the administration of inhaled anesthetic gases combined with intravenous drugs.

LBP patients showed changes in their neuromuscular activity, reduction in the lumbar muscle flexibility, and alteration of the biomechanical properties of the lumbar muscles.

ELIGIBILITY:
Inclusion Criteria:

1. All women gave birth through a cesarean delivery.
2. All women either primiparous or multiparous have not had anaesthesia (epidural, spinal, or general) for at least one year prior to the last obstetric anaesthesia.
3. Their ages ranged from 18 to 35 years.
4. All participants had a body mass index (BMI) of not more than 30, and a waist-to-hip ratio of not more than 1.
5. Participants were assessed between the 6th week to the 12th week postnatal.
6. All participants were able to continue all assessment procedures.
7. They were medically stable.

Exclusion Criteria:

1. Women who delivered through vaginal delivery.
2. Women who delivered through cesarean delivery, but the used anaesthetic technique was the paramedian approach for either the epidural or spinal anaesthesia.
3. Women with urinary tract infections.
4. Women who were below 18 years old or above 35 years old.
5. Women who had a (BMI) above 30 or a waist-to-hip ratio above 1.
6. Women who did not continue all assessment procedures.
7. Women who had any specific low back pain as women who were diagnosed with lumbar disc prolapse, scoliosis, or spondylolisthesis.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Because this study is presented to the department of Physical Therapy for Women's Health to observe the changes after cesarean delivery and its relevant anaesthesia.
Study Population: Sixty-three women participated in this study and were recruited from South Valley University Teaching Hospitals, in Qena governorate, Egypt.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Lumbar paravertebral muscle frequency (tone) | Assessment will be done 6-12 weeks after the use of anaesthesia for Cesarean section by the MyotonPRO device
  Tone is a contractile property of a muscle which describes the resting muscle's resistance to passive and active stretch forces
Lumbar paravertebral muscle stiffness | Assessment will be done 6-12 weeks after the use of anaesthesia for Cesarean section by the MyotonPRO device
  Stiffness is a biomechanical property of a muscle and its connective tissue which refers to the tissue's resistance toward the deformation of external load

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iddrisu M, Khan ZH. Anesthesia for cesarean delivery: general or regional anesthesia-a systematic review. Ain-Shams Journal of Anesthesiology. 2021 Dec;13(1):1-7.
- [Background] Mhyre JM, Sultan P. General Anesthesia for Cesarean Delivery: Occasionally Essential but Best Avoided. Anesthesiology. 2019 Jun;130(6):864-866. doi: 10.1097/ALN.0000000000002708. No abstract available. PMID 30985305
- [Background] Lenhardt R. Body temperature regulation and anesthesia. Handb Clin Neurol. 2018;157:635-644. doi: 10.1016/B978-0-444-64074-1.00037-9. PMID 30459029
- [Background] Struzik A, Karamanidis K, Lorimer A, Keogh JWL, Gajewski J. Application of Leg, Vertical, and Joint Stiffness in Running Performance: A Literature Overview. Appl Bionics Biomech. 2021 Oct 21;2021:9914278. doi: 10.1155/2021/9914278. eCollection 2021. PMID 34721664
- [Background] Van Deun B, Hobbelen JSM, Cagnie B, Van Eetvelde B, Van Den Noortgate N, Cambier D. Reproducible Measurements of Muscle Characteristics Using the MyotonPRO Device: Comparison Between Individuals With and Without Paratonia. J Geriatr Phys Ther. 2018 Oct/Dec;41(4):194-203. doi: 10.1519/JPT.0000000000000119. PMID 28005829
- [Background] Sung, S., and Mahdy, H. (2021):
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Hamilton RI, Garden CLP, Brown SJ. Immediate effect of a spinal mobilisation intervention on muscle stiffness, tone and elasticity in subjects with lower back pain - A randomized cross-over trial. J Bodyw Mov Ther. 2022 Jan;29:60-67. doi: 10.1016/j.jbmt.2021.09.032. Epub 2021 Oct 9. PMID 35248290
- [Background] Lo WLA, Yu Q, Mao Y, Li W, Hu C, Li L. Lumbar muscles biomechanical characteristics in young people with chronic spinal pain. BMC Musculoskelet Disord. 2019 Nov 23;20(1):559. doi: 10.1186/s12891-019-2935-z. PMID 31759390